CLINICAL TRIAL: NCT05649696
Title: A Single Bolus R-SAK Prior to Primary PCI for ST-elevation Myocardial Infarction (OPTIMA-5): 1-Year Follow-up
Brief Title: Prolonged Clinical Follow-up of OPTIMA-5
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chunjian Li, Director of Cardiology, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 020
Record Dates: First submitted 2022-11-24; First posted 2022-12-14 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-02

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI)
Keywords: ST Elevation Myocardial Infarction; Recombinant Staphylokinase
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- r-SAK group (Experimental): intravenous injection of single bolus 5 mg r-SAK in 3min
  Interventions: Drug: Recombinant Staphylokinase
- normal saline group (Placebo Comparator): intravenous injection of 10ml saline in 3min, r-SAK and saline are the same in appearance
  Interventions: Drug: Normal Saline
- patients with coronary artery disease (No Intervention): 20 ml arterial blood samples and 5 ml venous blood samples were collected from patients before coronary angiography

INTERVENTIONS:
Drug: Recombinant Staphylokinase — Intravenous injection of r-SAK is administered within 10 minutes after diagnosis of acute ST-segment elevation myocardial infarction
  Arms: r-SAK group
Drug: Normal Saline — Intravenous injection of normal saline is administered within 10 minutes after diagnosis of acute ST-segment elevation myocardial infarction
  Arms: normal saline group

SUMMARY:
The OPTIMA-5 trial is a prospective, multi-center, randomized, patient blinded, controlled trial comparing a single bolus of half-dose recombinant staphylokinase (r-SAK) with normal saline (NS) in patients with ST-segment elevation myocardial infarction (STEMI) presenting ≤12 hours of symptom onset and expected to undergo primary percutaneous coronary intervention (PPCI) within 120 minutes. The results of OPTIMA-5 showed that a single bolus r-SAK prior to PPCI for STEMI improves infarct related artery (IRA) patency and reduces infarct size without increasing major bleeding. On this basis, this study was designed to investigate the effect of the novel reperfusion strategy on 1-year outcomes of patients with STEMI.

DETAILED DESCRIPTION:
Acute myocardial infarction (AMI) is one of the leading causes of death all over the world, and accounted for more than 100 thousand deaths in the US in 2019. Early PPCI reduces mortality in patients with STEMI. If PPCI cannot be performed within 120 minutes of presentation, guidelines recommend the use of thrombolytic therapy. However, it remains uncertain whether adjunctive thrombolytic therapy administered immediately prior to PPCI improves outcomes in patients undergoing the procedure within 120 minutes.

SAK is a fibrin specific fibrinolytic agent produced by Staphylococcus aureus that was first discovered in 1948. A recombinant form of SAK was approved by China Food and Drug Administration (CFDA) for treatment of patients with STEMI. It has been demonstrated that r-SAK is more potent than urokinase and recombinant streptokinase in rabbit models.

The OPTIMA-5 trial is an investigator-initiated, prospective, multi-center, randomized, patient blinded, controlled trial comparing a single bolus of half-dose r-SAK with NS in patients with STEMI presenting ≤12 hours of symptom onset and expected to undergo PPCI within 120 minutes. Between October 29, 2021 and August 14, 2022, 283 STEMI patients were screened in 8 centers in China and 200 were randomized to r-SAK group or control in a 1:1 ratio using a computer-generated randomization sequence.

On this basis, this study was aimed to conduct a 1-year follow-up study to further confirm the efficacy and safety of this novel reperfusion strategy for patients with STEMI.

ELIGIBILITY:
Arm 1 and 2 inclusion and exclusion criteria

Inclusion Criteria:

1. Age 18-75 years, weight ≥45 kg;
2. Diagnosed as STEMI (meeting the following two criteria simultaneously):

   i. Ischemic chest pain lasts ≥30 minutes; ii. Electrocardiogram indicates that ST-segment elevation ≥2 mm in 2 or more contiguous precordial leads or ≥1 mm in 2 or more peripheral leads;
3. Time from onset of persistent chest pain to randomization <12 hours;
4. Primary PCI expected to be performed within 120 minutes.

Exclusion Criteria:

1. Cardiogenic shock;
2. Active bleeding or at high risk of bleeding (including grade Ⅲ or Ⅳ retinopathy or retinal gastrointestinal or urinary tract hemorrhage within the past 1 month);
3. Ischemic stroke or TIA in the past 6 months;
4. History of hemorrhagic stroke;
5. Platelet count <100×109/L or hemoglobin <100 g/L;
6. Known intracranial aneurysm;
7. Severe trauma, surgery or head injury within 1 month;
8. Suspected aortic dissection or infective endocarditis;
9. Recent puncture with difficult hemostasis by compression (eg, visceral biopsy, compartment puncture);
10. Currently taking anticoagulants;
11. Poorly controlled hypertension ( ≥180/110 mmHg);
12. Hepatic or renal impairment (glutamic-pyruvic transaminase, glutamic oxalacetic transaminase, or γ -glutamyl transferase >2.5 times upper limit of normal value; creatinine >1.5 times upper limit of normal value);
13. Known allergy to r-SAK;
14. Pregnancy, lactation, or planning for pregnancy;
15. History of myocardial infarction or CABG;
16. Having taken antiplatelet drugs other than aspirin and ticagrelor, such as clopidogrel, prasugrel or cilostazol after the symptom onset;
17. Patients with other conditions that made them unsuitable to be recruited at the discretion of the investigators.

Arm 3 inclusion and exclusion criteria Inclusion criteria

1. Age ≥18, ≤75 years old, weight ≥45kg, gender is not limited；
2. Taking maintenance dose of aspirin and ticagrelor for more than 3 days, or taking loading dose of aspirin (300mg) and ticagrelor (180mg);
3. Inpatients with suspected coronary atherosclerotic heart disease scheduled for coronary angiography or interventional therapy.

Exclusion criteria

1. Patients who had received r-SAK thrombolytic therapy before;
2. Previous diagnosis of Staphylococcus aureus infection;
3. Patients who were participating in other clinical trials;
4. Other patients considered unsuitable for inclusion by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
MACE | Within 360 days
  A composite of all-cause death, reinfarction, unplanned target vessel revascularization, heart failure or cardiogenic shock, major ventricular arrhythmia

SECONDARY OUTCOMES:
Adverse cardiac and cerebrovascular events | Within 360 days
  Each of the above independent MACE events, cardiovascular death, cardiac mechanical complications and stroke.

OTHER OUTCOMES:
r-SAK antibody level in human serum | Day 90 ± 7, Day 180 ± 7, Day 360 ± 14
  Recombinant staphylokinase (r-SAK) antibody level in human serum
In-vitro thrombolysis rate | 60 minutes after In-vitro thrombolysis
  In-vitro thrombolysis rate
r-SAK activity before and after in-vitro thrombolysis | Immediately before in-vitro thrombolysis and 60 minutes after In-vitro thrombolysis
  r-SAK activity before and after in-vitro thrombolysis

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Changzhou Second People's Hospital, Changzhou
  - The second Affiliated Hospital of Dalian Medical University, Dalian
  - Huai 'an Second People's Hospital affiliated to Nanjing Medical University, Huai'an
  - Lianyungang First People's Hospital, Lianyungang
  - Taizhou People's Hospital, Taizhou
  - Affiliated Hospital of Jiangnan University, Wuxi
  - The Second Affiliated Hospital of Zhejiang University Medical College, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Correction to: Heart Disease and Stroke Statistics-2018 Update: A Report From the American Heart Association. Circulation. 2018 Mar 20;137(12):e493. doi: 10.1161/CIR.0000000000000573. No abstract available. PMID 29555722
- [Background] Heusch G, Libby P, Gersh B, Yellon D, Bohm M, Lopaschuk G, Opie L. Cardiovascular remodelling in coronary artery disease and heart failure. Lancet. 2014 May 31;383(9932):1933-43. doi: 10.1016/S0140-6736(14)60107-0. Epub 2014 May 13. PMID 24831770
- [Background] Agnoletti G, Cargnoni A, Agnoletti L, Di Marcello M, Balzarini P, Pasini E, Gitti G, Martina P, Ardesi R, Ferrari R. Experimental ischemic cardiomyopathy: insights into remodeling, physiological adaptation, and humoral response. Ann Clin Lab Sci. 2006 Summer;36(3):333-40. PMID 16951276
- [Background] Townsend N, Wilson L, Bhatnagar P, Wickramasinghe K, Rayner M, Nichols M. Cardiovascular disease in Europe: epidemiological update 2016. Eur Heart J. 2016 Nov 7;37(42):3232-3245. doi: 10.1093/eurheartj/ehw334. Epub 2016 Aug 14. No abstract available. PMID 27523477
- [Background] Collen D, Lijnen HR. Thrombolytic agents. Thromb Haemost. 2005 Apr;93(4):627-30. doi: 10.1160/TH04-11-0724. PMID 15841305
- [Background] Pulicherla KK, Kumar A, Gadupudi GS, Kotra SR, Rao KR. In vitro characterization of a multifunctional staphylokinase variant with reduced reocclusion, produced from salt inducible E. coli GJ1158. Biomed Res Int. 2013;2013:297305. doi: 10.1155/2013/297305. Epub 2013 Aug 13. PMID 23998121
- [Background] Ueshima S, Matsuo O. Development of new fibrinolytic agents. Curr Pharm Des. 2006;12(7):849-57. doi: 10.2174/138161206776056065. PMID 16515501
- [Background] Yamamoto J, Kawano M, Hashimoto M, Sasaki Y, Yamashita T, Taka T, Watanabe S, Giddings JC. Adjuvant effect of antibodies against von Willebrand Factor, fibrinogen, and fibronectin on staphylokinase-induced thrombolysis as measured using mural thrombi formed in rat mesenteric venules. Thromb Res. 2000 Mar 1;97(5):327-33. doi: 10.1016/s0049-3848(99)00184-x. PMID 10709908
- [Background] Szemraj J, Stankiewicz A, Rozmyslowicz-Szerminska W, Mogielnicki A, Gromotowicz A, Buczko W, Oszajca K, Bartkowiak J, Chabielska E. A new recombinant thrombolytic and antithrombotic agent with higher fibrin affinity - a staphylokinase variant. An in-vivo study. Thromb Haemost. 2007 Jun;97(6):1037-45. doi: 10.1160/th06-10-0562. PMID 17549308
- [Background] Vakili B, Nezafat N, Negahdaripour M, Yari M, Zare B, Ghasemi Y. Staphylokinase Enzyme: An Overview of Structure, Function and Engineered Forms. Curr Pharm Biotechnol. 2017;18(13):1026-1037. doi: 10.2174/1389201019666180209121323. PMID 29424308
- [Background] Li CJ, Huang J, Yang ZJ, Cao KJ. Thrombolytic efficacy of native recombinant staphylokinase on femoral artery thrombus of rabbits. Acta Pharmacol Sin. 2007 Jan;28(1):58-65. doi: 10.1111/j.1745-7254.2007.00455.x. PMID 17184583
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). Glob Heart. 2018 Dec;13(4):305-338. doi: 10.1016/j.gheart.2018.08.004. Epub 2018 Aug 25. No abstract available. PMID 30154043
- [Background] Cutlip DE, Windecker S, Mehran R, Boam A, Cohen DJ, van Es GA, Steg PG, Morel MA, Mauri L, Vranckx P, McFadden E, Lansky A, Hamon M, Krucoff MW, Serruys PW; Academic Research Consortium. Clinical end points in coronary stent trials: a case for standardized definitions. Circulation. 2007 May 1;115(17):2344-51. doi: 10.1161/CIRCULATIONAHA.106.685313. PMID 17470709
- [Background] Halvorsen S, Storey RF, Rocca B, Sibbing D, Ten Berg J, Grove EL, Weiss TW, Collet JP, Andreotti F, Gulba DC, Lip GYH, Husted S, Vilahur G, Morais J, Verheugt FWA, Lanas A, Al-Shahi Salman R, Steg PG, Huber K; ESC Working Group on Thrombosis. Management of antithrombotic therapy after bleeding in patients with coronary artery disease and/or atrial fibrillation: expert consensus paper of the European Society of Cardiology Working Group on Thrombosis. Eur Heart J. 2017 May 14;38(19):1455-1462. doi: 10.1093/eurheartj/ehw454. No abstract available. PMID 27789570
- See also: OPTIMA-5 — https://clinicaltrials.gov/ct2/show/NCT05023681?term=NCT05023681&draw=2&rank=1